CLINICAL TRIAL: NCT03654508
Title: Pharmacogenetics Use For Further Treatment Improvement in childreN
Acronym: PUFFIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Lung Foundation (Unknown)
Responsible Party: Principal Investigator, Prof. dr. A.H. Maitland-van der Zee, Prof. dr. A.H. Maitland-van der Zee, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL63849.018.17
Record Dates: First submitted 2018-05-14; First posted 2018-08-31 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Asthma in Children
Keywords: long-acting beta2-agonist; pharmacogenetics

STUDY DESIGN:
Intervention Model Description: multicentre, double-blind, precision medicine, randomized trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADRB2-genotype guided treatment arm (Active Comparator): In the genotype-stratified arm, children will be treated based on their ADRB2 genotype. Children homozygous for the risk variant Arg16 and heterozygotes (Arg16Gly) will be treated with doubling dosages of their ICS. Children homozygous for the wild type allele (Gly16Gly) will receive LABA.
  Interventions: Genetic: ADRB2-genotype guided treatment
- Control arm (Active Comparator): In the control arm, genotyping will be performed for retrospective analysis, but the genotype information will not be used to guide treatment. Children in this study arm will proceed randomisation between doubling ICS dosage (n=75) or LABA treatment (n=75), the two most commonly preferred add-on options among paediatric pulmonologists in the Netherlands. The investigators choose to randomize between both treatments options, since international guidelines do not agree on the preferred treatment option.
  Interventions: Other: Randomisation

INTERVENTIONS:
Genetic: ADRB2-genotype guided treatment — This intervention assesses whether ADRB2 genotype-guided treatment leads to better asthma control after 3 months compared to usual care in children who are uncontrolled despite adherent and adequate use of ICS.
  Arms: ADRB2-genotype guided treatment arm
Other: Randomisation — In the control arm, children will be randomised over double dose ICS or ICS+LABA instead of treatment according to their genotype.
  Arms: Control arm

SUMMARY:
There is large heterogeneity in treatment response to asthma medication and a one-size fits all approach based on current guidelines might not fit all children with asthma. It is expected that children with one or more variant alleles (Arg16Arg and Arg16Gly) within the beta2 adrenergic receptor (ADRB2) gene coding for the beta2-receptor have a higher risk to poorly respond to long-acting beta2-agonists (LABA) comparing to the Gly16Gly wildtype.

Aims To study whether ADRB2 genotype-guided treatment will lead to improvement in asthma control in children with uncontrolled asthma on inhaled corticosteroids compared with usual care.

Design A multicentre, double-blind, precision medicine, randomized trial will be carried out within 20 Dutch hospitals. 310 asthmatic children (6-17 years of age) not well controlled on a low dose of inhaled corticosteroids (ICS) will be included and randomized over a genotype-guided and a non-genotype-guided(control) arm. In the genotype-guided arm children with Arg16Arg and Arg16Gly will be treated with double dosages of ICS and with the Gly16Gly wildtype with add on LABA. In the control arm children will be randomized over both treatment options. Lung function measurements, questionnaires focussing on asthma control (ACT/c-ACT) and quality of life, will be obtained in three visits within 6 months. The primary outcome will be improvement in asthma control based on repeated measurement analysis of c-ACT or ACT scores in the first three months of the trial. Additional cost effectiveness studies will be performed.

Conclusion Currently, pharmacogenetics is not used in paediatric asthmas. This trial may pave the way to implement promising results for genotype-guided treatment in paediatric asthma in clinical practice.

DETAILED DESCRIPTION:
Study design: national, multi-centre, double-blind randomized controlled trial

Duration: 6 months, with 3 visits in the hospitals (at t=0, t=3 months and t=6 months)

Setting: Patients are recruited at out-patient asthma clinics in secondary and tertiary care hospitals in the Netherlands.

Description: Three hundred ten children (6 to 17 years of age) with a doctor's diagnosis of asthma and uncontrolled asthma symptoms despite adherent and adequate use of ICS for at least three months (step 2 asthma treatment) will be recruited by secondary and tertiary care centers in the Netherlands. All participants are eligible for step-up asthma treatment (from step 2 to step 3) as assessed by the treating paediatrician/paediatric pulmonologist. Participants will be randomized to a genotype-guided treatment arm (n=155) or to a usual care, non-genotype guided arm (n=155) and followed for 6 months.

Genotyping before start treatment During the baseline visit in the hospital, clinical data and biological samples (including a DNA sample) will be collected. Upon this visit, the DNA sample will be send to the Clinical Chemistry department of the Erasmus MC (Head: Prof. R. van Schaik) to perform genotyping of the ADRB2 gene within one week. The treating physician will adapt the treatment regime of the participant based on the treatment advice of the study coordinator (Table 1). For the children in the genotype-arm, this will be based on the genotype. The treating physician will not know (be blinded) whether the treatment advice was based on the genotype (intervention arm) or based on randomization (control arm). The participant will be followed for 6 months. If the participant is still uncontrolled at t=3 months, treatment will be adapted. All children will be genotyped, in order to assess the influence of the genotype on treatment outcome in the usual arm group retrospectively. The children should use the same inhalation device during the study to avoid confusion on how they should inhale their medication.

Furthermore, to test the hypothesis it is necessary to include enough children in the control group with Arg16Arg or Arg16Gly to be treated with LABA. The amount of children treated with LABA and ICS should be equal in the control group. Therefore children are randomized in the control group over doubling ICS (n=77) and adding LABA (n=77). This will lead to an estimated number of children with Arg16Arg or Arg16Gly of 51 who will get LABA add on. In this way the power is high enough to determine the effectivity of both treatment options in the three genotypes. The investigators find it important to define effectivity next to the question whether genotyping benefits children with asthma. In the control group DNA samples will be obtained for retrospective analysis.

It is safe to randomise the children again who are randomised within the control arm, because treatment with a double dose of ICS and adding a LABA are both standard of care. A Cochrane review from 2009 has shown that both treatments have proven to be equally effective in both children and adults Randomisation in the control arm is important because it would be futile if the children in this arm would be treated with the same therapy by accident. Randomisation is necessary to make the trial as small and effective as possible. At this moment physicians do not have the tools to determine which therapy is the best for every child. This is why the investigators think it is correct to randomise in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Doctor's diagnosis of asthma (ever) based on patient history, FEV1 reversibility ≥ 12% and/or bronchial hyperresponsiveness
* Current asthma symptoms (based on ACT (≥12 years) or C-ACT (<12 years) score ≤ 19
* ICS use ≥ 3 months before inclusion (start dosage ICS, treatment step 2 according to childhood asthma guideline NVK, Table 3)
* Adequate inhalation technique (based on validated checklist score [21])
* Self-assessed good adherence to maintenance asthma treatment
* Understanding of Dutch language
* Internet access a home, willing to fill in internet questionnaires

Exclusion Criteria:

* Active smoking
* Congenital heart disease
* Serious lung disease other than asthma (Cystic Fibrosis, Primary Ciliary Dyskinesia, congenital lung disorders, severe immune disorders)
* LABA use in past 6 months
* Omalizumab use
* ICU admission in the previous year

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Asthma control based on (childhood-)Asthma Control Test scores in the first 3 months of the trial | 3 months
  Patients will fill in the (childhood-)Asthma Control Test at baseline, after 3 months [Range score: 0 - 27, 20 or more means asthma under control]

SECONDARY OUTCOMES:
Change in asthma control at t=6 months (childhood-)Asthma Control Test | 6 months
  Patients will fill in the (childhood-)Asthma Control Test at baseline after 6 months [Range score: 0 - 27, 20 or more means asthma under control]
Change in asthma-related school absences | 6 months
  Patients will fill in a questionnaire about asthma-related school absences [Minimum score 0 days, maximum score more than 10 days]
Change in therapy in t = 3 months | 3 months
  Patients will be questioned what kind of treatment they use at baseline visit, after three months
Time to reach asthma control (Asthma Control Test score ≥20) | 6 months
  Patients will fill in the (childhood-)Asthma Control Test at baseline, every month [Range score: 0 - 27, 20 or more means asthma under control]
Cost-effectiveness of ADRB2 genotype guided treatment measured by the Productivity Cost Questionnaire | 3 and 6 months
  Patients will fill in the Productivity Cost Questionnaire at 0, 3 and 6 months. The IPCQ measures:
  1. absenteeism (number of days missed from work in the 4 weeks due to illness) -- minimum is 0, maximum (in theory) is 28 days
  2. Presenteeism (productivity lost while at work due to illness) -- minimum is 0, maximum is 224 hours.
  In absenteeism, a lower number of days missed from work represent a better outcome; In presenteeism, a lower number of hours represent a better outcome For presenteeism the number of hours productivity loss is calculated by the following formula using data from the questionnaire.
  presenteeism = number of workdays affected by illness * (1-efficiencyscore/10)*working hours per workday.
  This results in a monetary value for productivity loss.
In-depth integrative -omics analysis | 0, 3 and 6 months
  Non-response to ICS treatment will be measured by analysing feces samples (microbiome) and nose swabs (epigenome). Nose swabs will be collected after 0, 3 and 6 months and feces after 1 month
Change in quality of life assessed by the Paediatric Asthma Quality of Life Questionnaire (PAQLQ) score | 0, 3 and 6 months
  Measured by the Pediatric Asthma-related Quality of Life Questionnaire (PAQLQ). Children are asked to think about how they have been during the previous week and to respond to each of the 32 questions on a 7-point scale (7 = not bothered at all -
  1 = extremely bothered). The overall PAQLQ score is the mean of all 23 responses and the individual domain scores are the means of the items in those domains. Subscales are summed.
Change in fatigue scores assessed by the PedsQL questionnaire | 0, 3 and 6 months
  Measured by the PedsQL questionnaire, a 23 item generic score scale consisting of physiological functioning, emotional functioning, social functioning and school functioning questions with multidimensional scales. Subscales are summed. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored.
change in FEV1 at t = 3 months | 0 and 3 months
  FEV1 will be measured at 0 and 3 months, change in FEV1 will be calculated.
change in FEV1 at t = 6 months | 0, 3 and 6 months
  FEV1 will be measured at t=0 and 6 months, change in FEV1 will be calculated
change in fraction of exhaled nitric oxide at t=3 months | 0 and 3 months
  Exhaled nitric oxide measures will be performed using the Niox Vero at t=0 and 3 months
change in fraction of exhaled nitric oxide at t=6 months | 0,3 and 6 months
  Exhaled nitric oxide measures will be performed using the Niox Vero at t=0. 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anke-Hilse Maitland-van der Zee, Prof. Dr., Principal Investigator — Academic Medical Center, Department of Respiratory Medicine
Locations (21):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Netherlands (19):
  - Nij Smellinghe, Drachten, Drenthe
  - Rijnstate, Arnhem, Gelderland
  - RadboudUMC, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Amphia ziekenhuis, Breda, North Brabant
  - Catharina ziekenhuis, Eindhoven, North Brabant
  - VUmc locatie Boelelaan, Amsterdam, North Holland
  - Academic Medical Center, Department of Respiratory Disease, Amsterdam-Zuidoost, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Sint Franciscus Gasthuis, Rotterdam, South Holland
  - Maasstadziekenhuis, Rotterdam, South Holland
  - Haga ziekenhuis, The Hague, South Holland
  - Medisch Spectrum Twente, Enschede, Twente
  - University Medical Center Groningen, Groningen
  - Martini ziekenhuis, Groningen
  - Tergooi ziekenhuis, Hilversum
- Kinderspital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03654508/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03654508/SAP_003.pdf